CLINICAL TRIAL: NCT00692549
Title: Ultrasound-Guided Peripheral Intravenous Cannulation in Emergency Department Patients With Difficult IV Access: a Randomized Trial.
Brief Title: Ultrasound Guidance for Intravenous Cannulation in Emergency Department Patients.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: John C. Stein MD, University of California, San Francisco
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RandomizedIVUS
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2008-06-06 (Estimated); Status verified 2008-06

CONDITIONS: Difficult IV Access
Keywords: ultrasound; iv access; Patients with difficult iv access in emergency departments.
MeSH Terms: interventions — Ultrasonography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ultrasound (Experimental): use of ultrasound
  Interventions: Device: ultrasound
- no ultrasound (No Intervention): no ultrasound

INTERVENTIONS:
Device: ultrasound
  Arms: Ultrasound

SUMMARY:
A randomized trial of the use of ultrasound by emergency physicians in the placement of intravenous catheters in emergency patients who are found to have difficult intravenous access (defined as two failed attempts by nursing staff).

ELIGIBILITY:
Inclusion Criteria:

* patients requiring an IV in the emergency department and who have two failed attempts by nursing staff

Exclusion Criteria:

* emergent need for IV access

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2005-06; Primary Completion 2005-08 (Actual); Study Completion 2005-08 (Actual)

PRIMARY OUTCOMES:
Number of IV Attempts

SECONDARY OUTCOMES:
Time to placement of IV catheter

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, San Francisco, California, United States